CLINICAL TRIAL: NCT07320430
Title: Comparative Study Between the Efficacy and Safety of Different Sclerosing Agents Used in Treatment of Low-Flow Vascular Malformation
Brief Title: Comparative Study Between Sclerosing Agents Used in Treatment of Vascular Malformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD15/2024
Record Dates: First submitted 2025-06-15; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-06

CONDITIONS: Vascular Malformation
Keywords: low-flow; sclerosing; vascular malformation
MeSH Terms: conditions — Vascular Malformations | interventions — Sclerotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- first group(Ethanol) (Active Comparator): * 25 patients receiving Ethanol 99.8% with maximum dose 1ml/kg/session
  * sclerotherapy with intralesional injection of ethanol for treatment of low-flow vascular malformation.
  Interventions: Procedure: sclerotherapy with intralesional injection of Ethanol for treatment of low-flow vascular malformatio
- second group(Bleomycin) (Active Comparator): 25 patients receiving bleomycin (15 U per bottle) will be reconstituted with 10 mL of normal saline to a final concentration of 1.5 U/ML, then 4ml will be foamed with 6ml human albumin.
  sclerotherapy with intralesional injection of bleomycin for treatment of low-flow vascular malformation.
  Interventions: Procedure: Sclerotherapy with intralesional bleomycin injection
- third group(Polidocanol) (Active Comparator): 25 patients receiving Polidocanol 3% which will be foamed 1ml+4ml air to a maximum dose of 15 ml /session.
  Interventions: Procedure: Sclerotherapy with intralesional injection of polidocanol

INTERVENTIONS:
Procedure: sclerotherapy with intralesional injection of Ethanol for treatment of low-flow vascular malformatio — First group will receive Ethanol. patients will be lying flat supine or prone according to the anatomical site of the lesion, US guided puncture of the vascular malformation (VM) using 21gauge butterfly needle under local, regional or light general anaesthesia according to the topography of the lesion and patient's age, when flow seen, contrast is used to confirm correct access, visualization of the vascular channels and any connection with arterial or deep venous system.
  injection of the sclerosing agent(Ethanol 99.8% with maximum dose 1ml/kg/session ) under fluoroscopy showing contrast displacement.
  After injection, DSA to allow visualization of negative or reduced dye filling, needle will be removed.
  compression will not be done for this group for fear of complications ( post operative pain- skin gangrene)
  Arms: first group(Ethanol)
Procedure: Sclerotherapy with intralesional bleomycin injection — second group will receive bleomycin. patients will be lying flat supine or prone according to the anatomical site of the lesion, US guided puncture of the vascular malformation (VM) using 21gauge butterfly needle under local, regional or light general anaesthesia according to the topography of the lesion and patient's age, when flow seen, contrast is used to confirm correct access, visualization of the vascular channels and any connection with arterial or deep venous system, injection of the sclerosing agent: bleomycin (15 U per bottle) will be reconstituted with 10 mL of normal saline to a final concentration of 1.5 U/ML, then 4ml will be foamed with 6ml human albumin, under fluoroscopy showing contrast displacement.
  After injection, DSA to allow visualization of negative or reduced dye filling, needle will be removed, then compression with bandage will be done .
  Arms: second group(Bleomycin)
Procedure: Sclerotherapy with intralesional injection of polidocanol — Third group will receive polidocanol. patients will be lying flat supine or prone according to the anatomical site of the lesion, torniquet is applied over the draining vein , US guided puncture of the VM using 21gauge butterfly needle under local, regional or light general anaesthesia according to the topography of the lesion and patient's age, when flow seen, contrast is used to confirm correct access, visualization of the vascular channels and any connection with arterial or deep venous system, injection of the sclerosing agent under fluoroscopy showing contrast displacement.
  polidocanol 3% will be foamed 1ml+4ml air to a maximum dose of 15 ml /session. After injection DSA to DSA to allow visualization of negative or reduced dye filling, needle will be removed, then compression with bandage .
  Arms: third group(Polidocanol)

SUMMARY:
This study aims to Compare the Efficacy and Safety of Different sclerosing Agents Used in Treatment of Low-Flow Vascular Malformation

DETAILED DESCRIPTION:
This study aims to Compare the Efficacy and Safety of Different sclerosing Agents Used in Treatment of Low-Flow Vascular Malformation.

Study Population: Patients with low -flow vascular malformations who visit Ain Shams University hospitals outpatient clinic.

* Type of Study: Randomized Controlled Clinical Trial.
* Study Setting: Ain Shams University hospitals.
* Study Period: 18 months.
* Sample Size: 75 patients.
* Sampling Method: Convenient sample, divided into three equal groups by closed enveloped method.

  * First group will receive ethanol, second group will receive bleomycin, and third group will receive polidocanol.

    * Study procedure: patients will be lying flat supine or prone according to the anatomical site of the lesion, torniquet is applied over the draining vein , US guided puncture of the VM using 21gauge butterfly needle under local, regional or light general anaesthesia according to the topography of the lesion and patient's age, when flow seen, contrast is used to confirm correct access, visualization of the vascular channels and any connection with arterial or deep venous system, injection of the sclerosing agent under fluoroscopy showing contrast displacement.
  * Ethanol 99.8% with maximum dose 1ml/kg/session, bleomycin (15 U per bottle) will be reconstituted with 10 mL of normal saline to a final concentration of 1.5 U/ML, then 4ml will be foamed with 6ml human albumin, polidocanol 3% will be foamed 1ml+4ml air to a maximum dose of 15 ml /session.
  * First group will receive ethanol, second group will receive bleomycin, and third group will receive polidocanol.
  * After injection, DSA to allow visualization of negative or reduced dye filling, needle will be removed, then compression with bandage except for ethanol group, with mean procedure time about 20 minutes

    * Medications:
  * Pre-operative: Prophylactic dose of anticoagulation will be given 5 days before operation for those with elevated D-dimer and will be continued for ten days post-operative.
  * Intraoperative: Each patient will receive an injection of 0.5 mg/kg of corticosteroids during the procedure.
  * Post-operative: PPI, oral corticosteroids- prednisolone 20mg once/day- for 5 days, anti-oedematous measures, and will be prescribed paracetamol tablets after the procedure.

    * Follow up:

The investigators will follow those patients clinically, and radiologically (follow up US&MRI selectively).

patients will be followed up few hours after operation, 2-4 weeks later between sessions, decision to continue the treatment or not will be made with the patient on the basis of the clinical efficacy. At the end of the treatment, patients will be followed up in a non-standardised manner up to 18 months, usually 1-3 months after the last session. When a consultation was not possible, telephone contact will be made with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schobinger stage II, III low- flow vascular malformation.
* Lesion affecting Patients trunk and extremity..
* Patient accepting the risk of the procedure and sign the detailed informed - consent, and in case of children-age less than18 years old- the consent will be signed by the parents

Exclusion Criteria:

* Patient with high- flow vascular malformation.
* Patients with schobinger I and IV AVM.
* Lesion affecting face, head, and neck.
* Vascular tumours; haemangioma.
* Patient with hypersensitivity to embolic agents e.g., hypersensitivity to bleomycin.
* Patients with CKD and elevated serum creatinine level.
* Critically ill patients Including pulmonary diseases, insufficient cardiac and hepatorenal functions, systemic infection, haemorrhagic tendency.
* Patient who /or his parents don't accept the risk of our procedure and don't sign the detailed informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
cure rate | 3 months after the last procedure
  cure rate defined as:
  1. Complete cure as 100% lesion devascularization on DSA or US with complete resolution of initial symptoms and signs.
  2. partial cure has been established as devascularization of 50%-99% with complete or partial resolution.

SECONDARY OUTCOMES:
Rate of complications . | within1 months after the last procedure
  1-Rate of complications including( pain, skin rash, hyperpigmentation, hypersensitivity reaction, PE
patient satisfaction | within 1 month after last procedure.
  Level of patient's satisfaction expressed through 5-point Likert scale.
  Items included are:
  1. Post-Operative Pain Management .
  2. Cosmetic Improvement .
  3. Functional improvement .
  4. Communication with the investigator about the case (diagnosis& management).
  5. Follow up after intervention.
  Overall Lowest score (5)means worst outcome, while Overall highest score (25)means best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hagag, Lecturer, MD vascular surgery, Study Director — faculty of medicine Ain shams Univerisity; Amr N kamel, professor of vascular surgery, Study Director — faculty of medicine Ain shams Univerisity; Ayman A Mohamed, professor of vascular surgery, Study Director — faculty of medicine Ain shams Univerisity
Locations (1):
- Faculty of medicine Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All available demographic data, photos taken before, during and after procedures, results can be shared
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- Available data/document: Study Protocol — https://www.mediafire.com/file/szzzndzizgwklut/mohamed_talat_MD_protocol.docx/file
- Available data/document: Informed Consent Form — https://www.mediafire.com/file/i75sevydp2nuygr/consent-.docx/file
- Available data/document: Analytic Code — https://www.mediafire.com/file/5g7dd95o0kd399p/5-ponts_likert_scale_for_patient_satisfaction.docx/file